CLINICAL TRIAL: NCT04263636
Title: Introduction of a Modified Luminous Efficiency Function V(λ)' That Addresses Total Light Transmittance of Patients That Underwent Pseudophakic Presbyopic Corrections
Brief Title: Luminous Efficiency Function V(λ)' of Patients That Underwent Pseudophakic Presbyopic Corrections
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Associate Professor of Ophthalmology, Democritus University of Thrace
Other Study IDs: ES11/Th12/27-12-2019
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Presbyopia
Keywords: pseudophakic presbyopic correction; trifocal intraocular lens; light intensity; eye light transmittance; light efficiency function
MeSH Terms: conditions — Presbyopia | interventions — Phacoemulsification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients that underwent uneventful bilateral pseudophakic presbyopic correction with trifocal diffractive IOLs (PanOptix or PanOptix toric, Alcon Laboratories, Inc., Fort Worth, TX, USA)
  Interventions: Procedure: Phacoemulsification with bilateral trifocal diffractive IOLs
- Control group: Patients of similar age without cataract that their crystalline lens has not been replaced.

INTERVENTIONS:
Procedure: Phacoemulsification with bilateral trifocal diffractive IOLs — Uneventful bilateral pseudophakic presbyopic correction with trifocal diffractive IOLs
  Groups: Study group

SUMMARY:
Primary objective of this study is to construct and validate a modified luminous efficiency function that addresses the distinct total eye light transmittance of patients that underwent bilateral pseudophakic presbyopic correction with trifocal intraocular lenses (IOLs) implantations.

DETAILED DESCRIPTION:
Present study aims to identify in which degree multifocal IOLs modify eye light transmission and estimate the necessary task and environmental lighting adjustment in order to address lighting needs of patients following bilateral pseudophakic presbyopic corrections. Specifically, the aim of this study is to identify the minimum light intensity in which patients that underwent pseudophakic presbyopic correction with trifocal IOLs can reach their maximum visual acuity (measured when lights are at the 100% lighting level)

ELIGIBILITY:
Inclusion Criteria:

* age between 45 to 70 years

Exclusion Criteria:

* astigmatism >1.00 diopters
* glaucoma
* former incisional eye surgery
* corneal or fundus disease
* diabetes mellitus
* autoimmune diseases
* neurological or psychiatric diseases
* posterior capsule rupture or lens misalignment
* postoperative uncorrected bilateral distant visual acuity < 8/10.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Presbyopic patients that underwent pseudophakic presbyopic correction with bilateral trifocal intraocular lenses implantation
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Minimum light intensity | 6 months postoperatively
  Minimum light intensity in which participants reach their maximum critical visual acuity

SECONDARY OUTCOMES:
Critical Visual Acuity (CVA) | 6 months postoperatively
  The print size of the optotype line fulfilling this criterion: all of the following lines are read at a time that is 1.96 times the standard deviation over the average reading time of the larger preceding lines. In clinical practice, the CVA is the minimum VA that can be read with the maximum possible speed.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Associate Professor
Locations (1):
- University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

REFERENCES:
- [Derived] Labiris G, Panagiotopoulou EK, Taliantzis S, Perente A, Delibasis K, Doulos LT. Lighting Standards Revisited: Introduction of a Mathematical Model for the Assessment of the Impact of Illuminance on Visual Acuity. Clin Ophthalmol. 2021 Nov 28;15:4553-4564. doi: 10.2147/OPTH.S326139. eCollection 2021. PMID 34866900